CLINICAL TRIAL: NCT06620978
Title: Operative Hysteroscopy Without Anaesthesia: Impact of Different Distention Medium Pressure (Using Normal Saline) on Visibility, Feasibility and Patients' Discomfort
Brief Title: Impact of Different Saline Pressures During Hysteroscopy on Visibility, Feasibility and Patients' Discomfort
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assaf-Harofeh Medical Center (Other Government)
Responsible Party: Principal Investigator, Neta Eisenberg Kogan, Attending physician in the gynecology endoscopic unit, Assaf-Harofeh Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 134-24-ASF
Record Dates: First submitted 2024-09-27; First posted 2024-10-01 (Actual); Last update posted 2024-10-02 (Actual); Status verified 2024-10

CONDITIONS: Endometrial Polyps; Retained Products of Conception; Lysis of Intrauterine Adhesions; Removal of Retained Intrauterine Device
MeSH Terms: interventions — Anesthesia

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Low pressure (Active Comparator): Low pressure (100 mmHg) Saline medium during hysteroscopy.
  Interventions: Procedure: Low pressure: Operative hysteroscopy without anesthesia with normal Saline medium in low pressure..
- High pressure (Active Comparator): High pressure (150 mmHg) Saline medium during hysteroscopy.
  Interventions: Procedure: High pressure: Operative hysteroscopy without anesthesia with normal Saline medium in High pressure.

INTERVENTIONS:
Procedure: Low pressure: Operative hysteroscopy without anesthesia with normal Saline medium in low pressure.. — Low pressure: Operative hysteroscopy without anesthesia with normal Saline medium in low pressure..
  Operative hysteroscopy without anesthesia using normal Saline as medium with different pressure according to the arm allocated. The procedure is done for endometrial polyp removal, retained products of conception removal, intrauterine adhesyolisis and intrauterine device removal.
  Arms: Low pressure
Procedure: High pressure: Operative hysteroscopy without anesthesia with normal Saline medium in High pressure. — High pressure: Operative hysteroscopy without anesthesia with normal Saline medium at high pressure.
  Arms: High pressure

SUMMARY:
Hysteroscopy is a minimally invasive diagnostic and therapeutic procedure for various intrauterine conditions. It is performed with an optic device while entering liquid media to the uterus to allow visualization. Diagnostic procedures are often performed without anaesthesia (in the office setting) and operative procedures are performed either under general anaesthesia or without anaesthesia (in the office setting). It depends on the patients' characteristics and preferences, and surgical indications. 80%-100% of operative procedure without anesthesia can be successfully completed. The main reasons for inability to successfully complete operative hysteroscopy without anesthesia are patients' discomfort and limited visibility of the uterine cavity.

In the current study, the investigators will compare the use of two different pressure setting of the liquid media during operative hysteroscopy without anesthesia, with the aim of investigating the successful completion of the procedure and patient's discomfort, with the aim of determining the optimal pressure setting.

DETAILED DESCRIPTION:
Hysteroscopy is a minimally invasive diagnostic and therapeutic procedure for various intrauterine conditions such as endometrial polyps, myomas, intrauterine adhesions, and retained products of conception. While the diagnostic procedures are often performed without anaesthesia (in the office setting), the operative procedures are performed either under general anaesthesia in the operative room, or without anaesthesia (in the office setting), depending on the patients' characterises and preferences, and surgical indications. In general, operative hysteroscopy without anaesthesia is offered to patients willing to undergo an awake operative procedure who have relatively small intrauterine pathologies (such as endometrial polyps and retained products of conception up to1.5 cm in diameter), mild intrauterine adhesions, and for removal of retained intrauterine device. In this setting, 80% to 100% of operative procedure without anesthesia can be successfully completed. The main reasons for inability to successfully complete operative hysteroscopy without anesthesia are patients' discomfort and limited visibility of the uterine cavity.

During hysteroscopy, distention of the uterine cavity with a distention medium is required to allow for optimal visualization. The uterine distention is an essential component of hysteroscopy, because the uterine cavity is a potential space which is normally collapsed. The most common distention medium for diagnostic and operative hysteroscopy is 0.9% normal saline. When the procedure is performed without anesthesia (i.e., in the office setting), some of the discomfort perceived by the patient is caused by the distention of the cavity. Obviously, longer procedures and the use of higher pressure of the distention medium are associated with greater patients' discomfort. On the other hand, the use of higher pressure may allow for better visualization of the uterine cavity, which may contribute to higher success rates of operative hysteroscopy without anesthesia. However, the optimal normal saline pressure which allows for adequate visualization of the uterine cavity and successful completion of operative hysteroscopy without anesthesia with acceptable patients' discomfort has not been determined to date. Previous studies have described the use of intrauterine pressure of normal saline for operative hysteroscopy without anesthesia in the range of 80 mmHg up to 150 mmHg.

In the current study, the investigators will compare the use of two different pressure setting for normal saline during operative hysteroscopy without anesthesia, with the aim of investigating the successful completion of the procedure, the surgeons' impression and the patient's discomfort, with the aim of determining the optimal pressure setting for these procedures.

Participation in the study will be offered to patients referred for operative hysteroscopy without anesthesia in the office setting in the outpatient service of the division of minimally invasive gynecologic surgery at the Shamir medical center department of obstetrics and gynecology. The indication for the surgery, surgical technique and instrumentation, and pre- and postoperative follow up will be identical to the standard procedures performed in our department in these cases. Patients will sign the standard informed consent form for operative hysteroscopy. Participants will be randomly assigned into the low pressure or the high pressure groups. The surgeons and the patients will be blinded to the pressure setting which will be set up by the assisting nurse. Following the procedure, the surgeon will fill a questionnaire regarding the feasibility of the procedure and the uterine cavity visibility (appendix 1). The intraoperative pain will be determined using a Visual analog scale (VAS).

ELIGIBILITY:
Inclusion Criteria:

1. Women age >18 years
2. Willing to undergo operative hysteroscopy without anesthesia for

The following intrauterine findings:

A. Endometrial polyps <1.5 cm B. Retained products of conception <1.5 cm C. Lysis of intrauterine adhesions D. Removal of retained intrauterine device

Exclusion Criteria:

1. Contraindication for hysteroscopy including: suspected pregnancy, heavy concomitant vaginal bleeding, known genital tract malignancy, suspected concurrent genital tract infection.
2. Unable to sign informed consent
3. Unable to read/write Hebrew

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Female gender
Enrollment: 100 (Estimated)
Dates: Start 2024-11-01 (Estimated); Primary Completion 2025-09-01 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
To compare the rate of successful completion rate of operative hysteroscopy without anesthesia using low pressure (100 mmHg) versus high pressure (150 mmHg) normal saline for distention medium. | The questionnaire will be filled immediately after the procedure.
  The feasibility and success of the procedure would be evaluated by the surgeon using a questionnaire.
Feasibility and uterine cavity visibility of operative hysteroscopy without anesthesia using low versus high pressure normal saline for distention medium. | The questionnaire will be filled immediately after the procedure.
  Feasibility and uterine cavity visibility of operative hysteroscopy without anesthesia using low pressure (100 mmHg) versus high pressure (150 mmHg) normal saline for distention medium. The feasibility of the procedure would be evaluated by the surgeon using a questionnaire.

SECONDARY OUTCOMES:
Patients' discomfort during operative hysteroscopy without anesthesia using low versus high pressure normal saline for distention medium. | Visual Analog Scale (VAS) will be filled immediately after the procedure.
  Patients' discomfort during operative hysteroscopy without anesthesia using low pressure (100 mmHg) versus high pressure (150 mmHg) normal saline for distention medium measured by VAS.

CONTACTS AND LOCATIONS:
Overall Officials: Neta Eisenberg Kogan, Principal Investigator — Assaf-Harofeh Medical Center

IPD SHARING:
Plan to Share IPD: Yes
Data collected and summarized by excel shits will be shared
Supporting Information: CSR
Time Frame: data will be available once study is completed for an unlimited period
Access Criteria: Will be shared via appropriated publications for public use

REFERENCES:
- [Background] Shahid A, Pathak M, Gulumser C, Parker S, Palmer E, Saridogan E. Optimum uterine filling pressure for outpatient diagnostic hysteroscopy: a double-blind, randomized controlled trial. Reprod Biomed Online. 2014 Jan;28(1):86-91. doi: 10.1016/j.rbmo.2013.07.018. Epub 2013 Sep 14. PMID 24262433
- [Background] De Silva PM, Stevenson H, Smith PP, Justin Clark T. A Systematic Review of the Effect of Type, Pressure, and Temperature of the Distension Medium on Pain During Office Hysteroscopy. J Minim Invasive Gynecol. 2021 Jun;28(6):1148-1159.e2. doi: 10.1016/j.jmig.2021.01.003. Epub 2021 Jan 11. PMID 33444792
- [Background] Salazar CA, Isaacson KB. Office Operative Hysteroscopy: An Update. J Minim Invasive Gynecol. 2018 Feb;25(2):199-208. doi: 10.1016/j.jmig.2017.08.009. Epub 2017 Aug 10. PMID 28803811
- See also: Enter the website. Type "Hysteroscopy managing fluid and gas distending media". — http://www.uptodate.com